12/06/2020

EFFECTS OF ERECTOR SPINAE PLANE BLOCK ON SYMPATHECTOMY IN OFF PUMP CORONARY ARTERY BYPASS SURGERY

## **INFORMED CONSENT FORM**

| EFFECTS OF ERECTOR SPINAE PLANE BLOCK ON SYMPATHECTOMY IN OFF PUMP CORONARY ARTERY BYPASS SURGERY |
|---|
| Initials of Volunteer: |
| Volunteer Number: |

"You are invited to a scientific research. Before you make your decision, it is important that you understand what this research entails and why. Please read the information below carefully and discuss it with your primary care physician, family and friends if necessary. If there is anything unclear or if you need further explanation, ask us. Think thoroughly whether you want to participate in this experiment or not."

# 1. What is the purpose of this study?

Off-pump coronary artery bypass grafting (OPCABG) is a bypass method performed on the working heart. Pain is a frequently seen side effect experienced following this surgery. Erector spina plane block is our analgesia method that we routinely perform prior to the surgery to overcome this problem. In this method, analgesic medication is given via a needle in between the two superficial muscle groups (erector spina muscles) located in your back. We believe this method not only provides pain relief, but also is beneficial (dilating) on the vessels that will be used for bypassing the clogged vessels during the surgery. We aimed to measure some parameters in this routine procedure before and after performing the analgesic method with an ultrasound (imaging with sound waves).

# 2. What will be the procedure performed on me?

In the pre-operative recovery room, an anesthesiology specialist will put on a lubricating gel on your thorax and perform imaging with an ultrasound. You won't feel any discomfort or pain during this imaging. The diameters of the vessels that might be used during your surgery for bypassing will be recorded via this imaging technique. Following this, our routine erector spina plane block will be performed where an analgesic medication will be given by an injection between the two superficial muscle groups on your back. Lastly, the vessel diameters on your thorax will again be recorded by an ultrasound with the help of the lubricating gel. The gel will be wiped off after imaging and you will be taken into the operating room.

# 3. What should I do if I join this research?

You don't need to do anything.

4. How long will the research take and how many volunteers will there be?

The research will last 2-3 months and there will be 25 volunteers.

5. Are there any side effects of the procedures on this research? What will happen if I develop these side effects?

No side effects are expected.

# 6. Who will meet the expenses that may arise from the medications, labs and exams? Will I need to pay anything?

There will be no payments for you or your social security institution.

- 6. Will the volunteers in this research be insured? No.
- 7. Will my participation in this study, my medical and personal information be confidential? Who will see these informations?

Your personal information won't be recorded. Your medical information will only be available to the researcher in charge and the associates.

- **8. Will this research be approved by an official authority?** Yes. It will be approved by the Koc University Ethical Committee.
- Whom can I contact if I need additional information or if there is a related emergency?

To acquire more information on the study or to consult on any side effects that may arise during the treatment, you may see your doctor. For more information, you can see Dr. Kamil DARCIN directly or reach him at 05055895099.

#### (Participiant's/Patient's Declaration)

Darticinant

It was stated that a medical research will be carried out in the Department of Anesthesiology and Reanimation at Koç University Faculty of Medicine and the above information about this research was conveyed to me. After this debriefing I was invited to participate in such research as "participant". If I participate in this research, I believe that the confidentiality of my information, that should stay between me and the physician, will be approached with great care and respect during this research. I was given sufficient reassurance that my personal information will be protected with utmost care during the use of research results for educational and scientific purposes. I can withdraw from the research without showing any reason during the execution of the project. (However, I am aware that it would be appropriate for me to notify in advance that I will withdraw from the research in order not to leave the researchers in a difficult situation.) I can also be excluded from the research by the researcher, provided that my medical condition is not harmed. I do not assume any monetary responsibility for the expenditures for the research. I will not receive a payment. Necessary assurance was provided that any medical intervention would be provided if any health problems that may arise from the research application, whether direct or indirect, occur. (I will not be under a monetary burden regarding these medical interventions.) I do not have to participate in this research and may not participate if I choose to do so. I have not encountered compelling behavior to participate in the research. I also know that if I refuse to participate, this will not harm my medical care and my relationship with the physician. I understand all the explanations made to me in detail. I decided to take part in this research project mentioned as a "participant" (subject) after a certain period of consideration on my own. I accept the invitation on this matter with great satisfaction and volunteerism. A copy of this signed form will be given to me.

Dhycician

| raiticipant | Pilysiciali |
|----------------|----------------|
| Name, Surname: | Name, Surname: |
| Address: | Address: |
| Phone: | Phone: |
| Signature | Signature |
| Witness | |
| Name, Surname: | |
| Adress: | |
| Signature: | |